CLINICAL TRIAL: NCT04090983
Title: Group-Based Cognitive-Behavioral Therapy for Adults With Attention-Deficit/Hyperactivity Disorder Inattentive Presentation: Randomized Controlled Trial
Brief Title: Cognitive-Behavioral Therapy for Adults With Attention-Deficit/Hyperactivity Disorder Inattentive Presentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Benjamin Bohman, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KI-2019-02444
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: ADHD Predominantly Inattentive Type
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-behavioral therapy (Hesslinger protocol) (Active Comparator)
  Interventions: Behavioral: Cognitive-behavioral therapy (Hesslinger protocol)
- Cognitive-behavioral therapy (CADDI protocol) (Experimental)
  Interventions: Behavioral: Cognitive-behavioral therapy (CADDI protocol)

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy (Hesslinger protocol) — Cognitive-behavioral therapy in a group format focusing on improving symptoms of ADHD, specifically by using skills in counteracting hyperactivity and impulsiveness, and promoting mindful awareness.
  Arms: Cognitive-behavioral therapy (Hesslinger protocol)
Behavioral: Cognitive-behavioral therapy (CADDI protocol) — Cognitive-behavioral therapy in a group format focusing on improving inattentive symptoms of ADHD, specifically by using skills in organizing, executing, and completing activity, and promoting mindful awareness.
  Arms: Cognitive-behavioral therapy (CADDI protocol)

SUMMARY:
Using a randomized controlled design, standard treatment of group cognitive-behavioral therapy (CBT) according to the Hesslinger protocol is compared to a newly developed group treatment specifically designed for adult patients with ADHD inattentive presentation (ADHD-I) called CBT for ADHD-I (CADDI). Research setting is psychiatric outpatient clinics. Research hypotheses include: 1. The CADDI protocol is more effective than standard treatment in terms of behavioral activation, procrastination, depressive symptoms, functional impairment, and quality of life, 2. Is equally effective in terms of ADHD symptoms, 3. Is more appreciated and tolerable, and 4. Outcome is mediated by mindful awareness. Effects are followed up at 6 and 12 months post treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Principal diagnosis of ADHD inattentive presentation
2. 18 years of age or older
3. If on medication, it needs to be well-established since three months, and
4. Prior psycho-educational intervention

Exclusion Criteria:

1. Intellectual impairment
2. Substance use disorder
3. Difficulties in adherence to medical or other treatment
4. Social and/or psychiatric problems to such an extent that they prevent focusing on treatment, or
5. Simultaneous psychological treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Behavioral Activation for Depression Scale | 14 weeks
  Total score 0-150; higher scores represent increased activation
Pure Procrastination Scale | 14 weeks
  Total score 12-60; higher scores represent more procrastination

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Bohman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Psychiatry Centre Södertälje, Södertälje, Stockholm County, Sweden